CLINICAL TRIAL: NCT03877263
Title: Comparing Specimen Collection Techniques to Screen for Sexually Transmitted Infections in Pregnant Women: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution and study was not transferred to anyone else.
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1297556
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Sexually Transmitted Diseases
Keywords: Chlamydia Trachomatis; Neisseria gonorrhoeae
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Masking Description: Patients agreeing to participate in the study will be randomized by visit into a study group in a 1:1 fashion. Patients who participate during both their initial and third trimester (of pregnancy) will be randomized twice to a study group.
  The randomization allocation schedule will be developed by biostatisticians from the OhioHealth Research & Innovation Institute (OHRI), and will be hidden from the investigator until directly prior to enrollment to prevent bias. The clinical research coordinator will reveal the randomization allocation once patient is consented and enrolled into the study.
  Due to the nature of the study, we cannot completed mask the investigator from the study group while taking the vaginal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OB/GYN physician-collected vaginal swab (Other): Patients assigned to the physician-collected vaginal swab group will have their Vaginal swab for detection of STI collected by their obstetrics and gynecology (OB/GYN) physician.
  The vaginal swabs will be collected first for all patients, to avoid any swab contact with lubricant. As standard of care, the physician will collect Endocervical swab for detection of STI for this group.
  Interventions: Diagnostic Test: Endocervical swab for detection of STI; Diagnostic Test: Vaginal swab for detection of STI
- Patient-collected vaginal swab (Other): Patients assigned to the patient-collected vaginal swab group will self-collect the Vaginal swab for detection of sexually transmitted infection (STI). Patients who self-collect will receive instructions from their OB/GYN physician and in paper form.
  The vaginal swabs will be collected first for all patients, to avoid any swab contact with lubricant. As standard of care, the physician will collect Endocervical swab for detection of STI for this group.
  Interventions: Diagnostic Test: Endocervical swab for detection of STI; Diagnostic Test: Vaginal swab for detection of STI

INTERVENTIONS:
Diagnostic Test: Endocervical swab for detection of STI — After we collect the samples, they will be evaluated using the Hologic APTIMA Chlamydia trachomatis and Neisseria gonorrhoeae assays.
Diagnostic Test: Vaginal swab for detection of STI — After we collect the samples, they will be evaluated using the Hologic APTIMA Chlamydia trachomatis and Neisseria gonorrhoeae assays.
  We will then compare the results from a vaginal vs. endocervical specimens within and between the groups

SUMMARY:
The purpose of this research study is to compare two specimen collection techniques (vaginal vs. endocervical swab) to screen for sexually transmitted infections in pregnant women. Either a physician or the patient may collect the vaginal specimen; the physician will collect the endocervical specimen during a standard-of-care pelvic exam. Each technique utilizes a specialized swab for specimen collection. We will used the Hologic Aptima C. trachomatis and N. gonorrhoeae detection assay to analyze both specimens.

We hypothesize that the results from the physician-collected vaginal specimen will have equivalent outcomes those from the physician-collected endocervical specimen. If the techniques are equivalent for detecting infection, there may be an opportunity for cost saving and increased patient satisfaction with the vaginal technique, especially using patient-collected vaginal specimen collection.

DETAILED DESCRIPTION:
Chlamydia trachomatis and Neisseria gonorrhoeae are the two most commonly reported infectious diseases in the United States. Their role in pregnancy-related comorbidities such as spontaneous abortion, preterm labor, chorioamnionitis, preterm premature rupture of membranes, and perinatal infection is complicated as data is conflicting. Many reports suggest increased risks of adverse pregnancy outcomes in the presence of C. trachomatis and N. gonorrhoeae infections. However, there are also several studies that have failed to demonstrate an increased risk. Despite conflicting reports, due to high prevalence of these infections and association with pregnancy-related co-morbidities, the Center for Disease Control (CDC) recommends screening for C. trachomatis and N. gonorrhoeae in high-risk populations at initiation of prenatal care, and again during the third trimester to ensure infections are treated quickly and resolved prior to birth.

In the non-pregnant female population, there are many ways to screen for C. trachomatis and N. gonorrhoeae pelvic infections, including bacterial culture, direct fluorescent antibody testing, deoxyribonucleic acid (DNA) probe, enzyme immunoassay, or ribonucleic acid (RNA) amplification. These various testing modalities can be applied to urine, or vaginal or endocervical samplings. RNA assays and DNA probes are currently the least expensive and most accurate way of screening, and are therefore the most routinely used.

At OhioHealth Doctors Hospital (DH) Women's Health Center, pregnant patients are screened for sexually transmitted infections (STI) using the Hologic Aptima Chlamydia trachomatis and the Neisseria gonorrhoeae assays, which are second generation nucleic acid amplification assays (NAATs). Samples are collected using the Hologic Aptima Unisex Specimen Collection Kit for Endocervical and Male Urethral Swab Specimens. These swabs are specifically designed for cervical swab collection techniques. Per standard of care at DH and CDC recommendations, patient endocervical swabs are collected at the patient's initial prenatal visit and during her third trimester appointment (approximately 36 week gestation) to test for infection.

In non-pregnant women, the vaginal specimen collection kit has been shown to be just as effective at detecting pelvic infections of C. trachomatis and N. gonorrhea using RNA assays. There are many benefits of adopting the use of a vaginal specimen collection kit, as compared to endocervical collection. Vaginal sampling can be performed without a speculum exam in asymptomatic women. In addition to being a less invasive test, the vaginal swab may reduce testing costs, by eliminating the use of collection tools (such as disposable speculums) that are required during an endocervical collection; avoiding the endocervical collection procedure may also reduce the overall office visit time. Additionally, patients could be instructed to collect a vaginal sample themselves. This may increase patient satisfaction, privacy, and comfort. In fact, several publications have reported patient preference for a self-collected vaginal swab vs. an endocervical swab.

Few studies have evaluated the used of vaginal or introital swabbing techniques for detection of infectious microorganisms during pregnancy, but the published data is favorable for the use of a vaginal swab. Thus, more data is needed to compare the use of vaginal vs. endocervical swabs to detect infections in pregnant women. The objective of this study is to compare detection of sexually transmitted infections in pregnant women by collecting samples using both the Hologic Aptima Vaginal Swab and the Unisex Specimen Collection Kit for Endocervical and Male Urethral Swab.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant & receiving prenatal care at Doctors Hospital Women's Health Center
2. ≥16 years old
3. Able to understand & consent to study participation
4. English speaking & reading; if minor assent form is required, the parent or guardian must also be English speaking & reading

Exclusion Criteria:

1. Females who are not pregnant.
2. <16 years old.
3. Not english speaking & reading; if minor assent form is required, the parent or guardian are not english speaking & reading

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Compare the physician-collected vaginal swab outcomes to those from the physician-collected endocervical swab. | 12 months
  Determine the rate of concordance for infection screening results between the physician collected vaginal and physician collected endocervical specimens in pregnant patients. Concordance will be defined as same results (whether positive or negative) on both methods.

SECONDARY OUTCOMES:
Assess the costs of medical supplies used during pelvic examinations. | 12 months
  Compare the costs of medical supplies used in endocervical vs vaginal sample collection techniques.

OTHER OUTCOMES:
Patient satisfaction following specimen collection. | 12 months
  We will describe patient satisfaction following specimen collection using a patient-collected vaginal swab, a physician-collected vaginal swab, or a physician-collected endocervical swab.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Topolnycky, DO, Study Chair — Attending Physician; Krista Jensen, DO, Principal Investigator — Resident Physician
Locations (1):
- OhioHealth Doctors Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be collected using study-specific data abstraction sheets/data collection tools (e.g., REDCap or Excel). Only institutional review board (IRB)-approved variables will be collected. Electronic files will be stored on a password-protected computer, and paper files will be stored in a secure facility with limited access (the offices of the OhioHealth Research Institute). Desktop or mobile computers used for research purposes will be password-protected and encrypted. Data transmitted over the internet or via email will be encrypted.
  All resulting data will be securely stored in electronic format according to OhioHealth policy; the data collection and storage processes will follow HIPAA guidelines in accordance to 45 Code of Federal Regulations (CFR) Part 160 & 164, to protect both confidentiality and privacy of each participant. All protected health information (PHI) data will be released or destroyed per institution protocol.